CLINICAL TRIAL: NCT07156227
Title: Phase I Trial of ATR Inhibitor Camonsertib Combined With Stereotactic Body Radiation Therapy for Recurrent Head and Neck Squamous Cell Carcinoma
Brief Title: Testing the Addition of an Anti-Cancer Drug, Camonsertib, to Radiation Therapy for Recurrent Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-06201; NCI-2025-06201 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10732 (Other: UPMC Hillman Cancer Center LAO); 10732 (Other: CTEP); UM1CA186690 (NIH)
Record Dates: First submitted 2025-09-04; First posted 2025-09-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Recurrent Paranasal Sinus Squamous Cell Carcinoma; Stage III Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage III Sinonasal Cancer AJCC v8; Stage IV Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage IVA Hypopharyngeal Carcinoma AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVA Lip and Oral Cavity Cancer AJCC v8; Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVA Sinonasal Cancer AJCC v8; Stage IVB Hypopharyngeal Carcinoma AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVB Lip and Oral Cavity Cancer AJCC v8; Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVB Sinonasal Cancer AJCC v8; Unresectable Head and Neck Squamous Cell Carcinoma; Unresectable Hypopharyngeal Squamous Cell Carcinoma; Unresectable Laryngeal Squamous Cell Carcinoma; Unresectable Oral Cavity Squamous Cell Carcinoma; Unresectable Oropharyngeal Squamous Cell Carcinoma; Unresectable Paranasal Sinus Squamous Cell Carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Carcinoma | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (camonsertib, SBRT) (Experimental): Patients undergo SBRT twice weekly, 2-3 days apart, for 4 or 5 fractions over 3 weeks. Patients receive camonsertib PO QD on the day of and the day after each radiation therapy treatment. Patients also undergo PET/CT or CT and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Camonsertib; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Camonsertib — Given PO
  Other Names: ATR Inhibitor RP-3500; RP 3500; RP-3500; RP3500
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of camonsertib in combination with stereotactic body radiation therapy in controlling disease in patients with head and neck squamous cell cancer that has come back after a period of improvement (recurrent) or that cannot be removed by surgery (unresectable). Camonsertib may stop the growth of tumor cells and may kill them by blocking some of the enzymes needed for cell growth. Stereotactic body radiation therapy is a type of external radiation therapy that uses special equipment to position a patient and precisely deliver radiation to tumors in the body (except the brain). The total dose of radiation is divided into smaller doses given over several days. This type of radiation therapy helps spare normal tissue. Giving camonsertib in combination with stereotactic body radiation therapy may help control disease in patients with recurrent or unresectable head and neck squamous cell cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of camonsertib with concurrent head and neck stereotactic body radiotherapy (SBRT) reirradiation for patients with recurrent head and neck squamous cell carcinoma (HNSCC).

II. To determine the recommended phase 2 dose (RP2D) of camonsertib in combination with concurrent SBRT in these patients.

SECONDARY OBJECTIVES:

I. To assess overall response rate within the radiation therapy field for patients treated with camonsertib and SBRT.

II. To assess progression-free survival (PFS) with camonsertib and SBRT in patients with recurrent or new primary HNSCC within a previously irradiated field.

EXPLORATORY OBJECTIVES:

I. To identify predictive biomarkers of response to camonsertib and SBRT, including, but not limited to genetic alterations of ATM and TP53, human papillomavirus (HPV) status, tumor mutational load, and circulating tumor deoxyribonucleic acid (DNA).

II. To characterize the pharmacokinetics (PK) of camonsertib.

OUTLINE: This is a dose-escalation study of camonsertib in combination with SBRT followed by a dose-expansion study.

Patients undergo SBRT twice weekly, 2-3 days apart, for 4 or 5 fractions over 3 weeks. Patients receive camonsertib orally (PO) once daily (QD) on the day of and the day after each radiation therapy treatment. Patients also undergo positron emission tomography (PET)/computed tomography (CT) or CT and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up at weeks 4, 5, 6, 7, 16, 29, 42, and 55.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed recurrent or metachronous (second primary) unresectable head and neck squamous cell carcinoma involving the oral cavity, oropharynx, larynx, hypopharynx, and/or paranasal sinus, or cervical lymphadenopathy with unknown primary. Core needle biopsy (preferably at least three 18-gauge cores) or incisional biopsy is preferred over fine needle aspiration (FNA) for diagnosis of recurrent disease or new primary head and neck squamous cell carcinoma to provide sufficient tumor tissue for correlative studies. Unresectable refers both to patients who have declined surgery and patients deemed unresectable by otolaryngology. This includes patients for whom curative resection is medically contraindicated and/or would be associated with excessive surgical risk (as deemed by the consulting otolaryngologist) or undue surgical morbidity (e.g., total glossectomy, laryngectomy, and/or major resection requiring free flap reconstruction)
* Patients must have recurrent disease within a previously irradiated area (radiotherapy to dose ≥ 30 gray [Gy]; in-field recurrence)
* Patients must have completed prior radiotherapy at least 6 months prior to enrollment. Due to safety concerns, reirradiation within less than 6 months to the head and neck is very rarely recommended per standard of care
* Patients must have measurable disease (at least one measurable lesion) as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Baseline imaging must include neck CT (preferably contrast-enhanced) and chest CT or skullbase to midthigh PET/CT (preferably with contrast-enhanced neck CT if diagnostic contrast-enhanced neck CT not available). Patients who have undergone surgery aside from biopsy may be included if gross disease is present within the surgical resection bed or at another site
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of camonsertib in combination with radiotherapy in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Leukocyte count ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or erythropoietin dependency (within 7 days of assessment)
* Serum bilirubin ≤ 1.5 × institutional upper limit of normal (ULN) (if total serum bilirubin > 1.5 × institutional ULN, then direct bilirubin must be < ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3 × institutional ULN
* Albumin > 2.5 mg/dL
* Glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m^2

  * GFR can be measured directly or estimated using the site's institutional standards
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Ability to take pills by mouth
* The effects of camonsertib on the developing human fetus are unknown. For this reason and because ATR inhibitors and radiation are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after completion of camonsertib administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1), with the exception of alopecia
* Patients who are receiving any other investigational agents for a current cancer diagnosis
* Patients with distant metastatic disease
* Patients who have received more than one prior course of head and neck radiotherapy
* Patients who have disease surrounding > 180 degrees of the carotid artery
* Patients with tumors invading the mandible or tumors with gross skin involvement (i.e., tumor ulceration through the skin)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to camonsertib or radiation
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because camonsertib is an ATR inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with camonsertib, breastfeeding should be discontinued if the mother is treated with camonsertib. These potential risks may also apply to other agents used in this study
* Patients diagnosed with scleroderma
* Concomitant use of strong CYP3A4/5 inhibitors and inducers, and strong P-gp and BCRP inhibitors

  * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-03-26 (Estimated); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | During dose escalation phase
  The safety and tolerability of camonsertib will be evaluated during the dose escalation phase. The frequency and percentage of AEs will be provided overall and by dose level for any grade and attribution as well as for grade 3 or greater AEs, at least possibly related to treatment.
Maximum tolerated dose (MTD) of camonsertib and concurrent stereotactic body radiation therapy (SBRT) reirradiation | During dose escalation phase
  The dose-escalation phase will utilize a Bayesian Optimal Interval Design to determine the MTD for combined camonsertib and SBRT.
Incidence of late toxicities (dose expansion phase) | Within 1 year of treatment initiation
  The proportions of total patients experiencing late toxicities will be estimated. The frequency and percentage of AEs will be provided overall and by dose level for any grade and attribution as well as for grade 3 or greater AEs, at least possibly related to treatment.

SECONDARY OUTCOMES:
Overall response rate | Up to 55 weeks
  Will be evaluated within the radiation therapy field. Overall response will be defined as a complete or partial response based on the Response Evaluation Criteria in Solid Tumors 1.1 criteria. The proportion of patients responding to the treatment regimen and corresponding 95% confidence interval estimates will be calculated.
Progression-free survival (PFS) | From the start of treatment regimen until documented local or distal failure or death from any cause, assessed up to 55 weeks
  PFS will be estimated using the method of Kaplan-Meier.

OTHER OUTCOMES:
Biomarkers of response | Up to 55 weeks
Pharmacokinetic data | Day 1: Pre, and 0.5, 1, 1.5, 2, 4, 6, and 8 hour post and Day 2: 24 hour after dose 1, pre-dose 2

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne M Mowery, Principal Investigator — UPMC Hillman Cancer Center LAO

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm